CLINICAL TRIAL: NCT03483480
Title: Randomized Controlled Trial of Non-Powered Negative Pressure Wound Therapy vs Open Technique for Pilonidal Disease
Brief Title: Non-Powered Negative Pressure Wound Therapy vs Open Technique for Pilonidal Disease
Acronym: NPWTvsOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The National Children's Hospital, Tallaght (Other)
Responsible Party: Principal Investigator, Yasir Bashir, Assistant Professor of Surgery, The National Children's Hospital, Tallaght
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-02
Record Dates: First submitted 2018-03-17; First posted 2018-03-30 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Pilonidal Disease; Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non powered-NPWT (Experimental)
  Interventions: Procedure: NPWT for Pilonidal Surgery
- Open Technique (Active Comparator)
  Interventions: Procedure: Excision of Pilonidal sinus with normal dressing

INTERVENTIONS:
Procedure: NPWT for Pilonidal Surgery — After excision of pilonidal sinus Non powered-NPWT will be applied to the area
  Arms: Non powered-NPWT
Procedure: Excision of Pilonidal sinus with normal dressing — After excision of pilonidal sinus normal dressing will be applied to the area of surgery
  Arms: Open Technique

SUMMARY:
Pilonidal Disease is disease of young patients with significant morbidity and is difficult to treat. Currently multiple methods are practiced for the treatment of the disease, two of them are preferred over others and practice extensively. First one involves excision of pilonidal sinus and dressings while the second one is excision of the pilonidal sinus with application of negative pressure wound therapy. None of these approaches is considered superior to the other, as not enough comparison studies of the two procedures have been done. In order to clarify this and find the best option for our patients, investigators are taking opportunity to compare these two modalities. If participants choose to participate in this study they will be randomly selected to one of these groups and the progress of wound healing will be monitored after surgery with the measurement of wound weekly and photographs. Investigators are hoping to find out which procedure is superior. This will allow investigators to provide the best treatment option for their patients in future.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient suffering from Pilonidal Disease willing to participate in study.

Exclusion Criteria:

* Patients below the age of 16 years (not able to consent).
* Not consenting to participate in study.
* Patient with less than 3 cm between inferior opening of sinus and anus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound healing | Wound will be assessed for healing at 1 week to 6 weeks
  Time between Surgery and complete healing when there is no further requirement to apply dressing

SECONDARY OUTCOMES:
VAS score (Visual Analogue Scale) | VAS for pain will be recorded at 1 week to 6 weeks at weekly intervals
  Pain score as scored by patients, VAS is an analogue scale is from 1 to 10, 1 being minimal discomfort to 10 being the worst pain in the life
Wound size ratio | Wound size ratio will be recorded at 1 week to 6 weeks at weekly intervals
  Healing as ratio of the initial wound
Time to resume daily activities | Assessment will be done at 1 week to 6 weeks at weekly intervals
  Time at which patient is able to do his/her daily household works
Recurrence | Patient will be assessed at 6 months from surgery
  Recurrence of disease at 6 months from surgery
Analgesia Requirement | Recording will be done at 1 week to 6 weeks at weekly intervals
  Requirement for analgesia will be recorded to make the pain analysis more robust

CONTACTS AND LOCATIONS:
Locations (1):
- Tallaght Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: data will be available on request for 3 months at publication of study
Access Criteria: Send email to Principal Investigator with query and information needed. Principal Investigator will reply as soon as possible and provide the information requested.